CLINICAL TRIAL: NCT02802111
Title: Change in Oxygen Consumption Following Inhalation of Albuterol in Comparison With Levalbuterol in Healthy Adult Volunteers
Brief Title: Change in Oxygen Consumption Following Inhalation Beta Agonists in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Patrick Ross, Associate Professor of Clinical Anesthesia and Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CCI-14-00101
Record Dates: First submitted 2016-06-10; First posted 2016-06-16 (Estimated); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Oxygen Consumption
Keywords: Beta Agonists; Asthma; Albuterol; Levalbuterol
MeSH Terms: conditions — Asthma | interventions — Albuterol; Levalbuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol 5 mg first, then levalbuterol 2.5 mg (Experimental): Patient receives albuterol 5 mg aerosolized first and then 4 hours or greater after receives levalbuterol 2.5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention.
  Interventions: Drug: Albuterol
- Levalbuterol 2.5 mg first, then albuterol 5 mg (Experimental): Patient receives levalbuterol 2.5 mg aerosolized first and then 4 hours or greater after receives albuterol 5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention.
  Interventions: Drug: Levalbuterol

INTERVENTIONS:
Drug: Albuterol — Patient receives albuterol 5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention.
  Arms: Albuterol 5 mg first, then levalbuterol 2.5 mg
Drug: Levalbuterol — Patient receives levalbuterol 2.5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention
  Arms: Levalbuterol 2.5 mg first, then albuterol 5 mg

SUMMARY:
Albuterol is the most commonly used β agonist to treat reversible lower airway obstruction. Albuterol contains a racemic mixture of two enantiomers. Levalbuterol contains the single R form enantiomer. Levalbuterol is frequently prescribed to limit cardiovascular toxicity. The investigators sought to examine the changes in oxygen consumption (V'O2) and Heart Rate (HR) following administration of albuterol and

DETAILED DESCRIPTION:
Inhaled β2 adrenoceptor agonists are frequently used to treat reversible lower airway obstruction, or to assist with mucociliary clearance. Albuterol remains the most commonly used β agonist and contains a racemic mixture of two enantiomers. The R enantiomer is the active moiety responsible for the bronchodilation, while the S enantiomer was initially thought to be inactive, although recent studies suggest otherwise. Levalbuterol contains the single R form enantiomer, and in clinical practice it is frequently prescribed not only because of its bronchodilator benefits, but to limit cardiovascular toxicity. Adverse cardiovascular effects remain the main dose-limiting factor for β2 agonists. The primary objective of the investigators study is to compare the change in oxygen consumption following albuterol to that of levalbuterol, in healthy adult volunteers. The investigators hypothesized there would be no clinically significant difference in V'O2 between the two drugs, if equal doses of the R-enantiomer were administered. Secondary objectives were to compare the changes in heart rate and other vital signs between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18 and 60 years

Exclusion Criteria:

* Coronary artery disease, history of intolerance to beta agonists

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Ross, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (5 Min of Drug)
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout (4 Hours)
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention (5 Min of Drug)
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 30 [19 to 40] | 34 [24 to 53] | 32 [19 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 0 | 0 | 0
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Consumption
Description: Oxygen consumption will be measured following for up to 60 minutes beta agonist aerosol
Time Frame: 0 to 60 minutes
Population: Healthy volunteers, median age 32 years. The population is 24 individuals they are randomized to which bronchodilator they received first. Half were randomized to Albuterol and half to levalbuterol but each subject received both medication. It is a matter of which they received first. There was a four hour wash out period between the first and second medication.
Measure: Median (Inter-Quartile Range); unit: mls/kg/min
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
Number analyzed (Participants) | 24 | 24
mls/kg/min | .28 [.15 to .36] | .27 [.19 to .35]

2. Secondary Outcome: Heart Rate
Description: Vital signs including heart rate will be measured for up to 60 minutes following beta agonist
Time Frame: 0 to 60 minutes
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
Number analyzed (Participants) | 24 | 24
beats per minute | 91 [84 to 103] | 93 [87 to 102]

ADVERSE EVENTS:
Time Frame: We observed the volunteers over 4 hours following use of either albuterol first or levalbuterol first then for another 4 hours following the second medication.
Description: We observed the volunteers over 4 hours following use of either albuterol first or levalbuterol first then for another 4 hours following the second medication. If there were an adverse event we would record it in the area for the first medication that they received. Overall there were no adverse events.
Groups:
- Albuterol 5 mg First, Then Levalbuterol 2.5 mg: Patient receives albuterol 5 mg aerosolized first and then 4 hours or greater after receives levalbuterol 2.5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention. Patients are observed for adverse events for 4 hours after second medication.
  Albuterol: Patient receives albuterol 5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention.
- Levalbuterol 2.5 mg First, Then Albuterol 5 mg: Patient receives levalbuterol 2.5 mg aerosolized first and then 4 hours or greater after receives albuterol 5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention. Patients are observed for adverse events for 4 hours after second medication.
  Levalbuterol: Patient receives levalbuterol 2.5 mg aerosolized. Oxygen consumption and vital signs are measured for 1 hour after intervention
Arm/Group | Albuterol 5 mg First, Then Levalbuterol 2.5 mg | Levalbuterol 2.5 mg First, Then Albuterol 5 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT02802111/Prot_SAP_000.pdf